CLINICAL TRIAL: NCT03438786
Title: Trans-inguinal Pre-peritoneal (TIPP) Hernioplasty Versus Lichtnestein's Technique in Inguinal Hernia Repair
Brief Title: Trans-inguinal Pre-peritoneal Hernioplasty Versus Lichtnestein's Technique in Inguinal Hernia Repair
Acronym: TIPP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamad Hamdy, Resident doctor at General surgery department, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: inguinal hernia
Record Dates: First submitted 2018-01-23; First posted 2018-02-20 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Intervention Model Description: patients will be randomized into two groups according to the surgical technique performed as follows :-
  * Group A: Patients undergoing TIPP hernioplasty
  * Group B: Patients undergoing lichtnestein's technique hernioplasty
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): Patients undergoing trans-inguinal pre-peritoneal (TIPP) hernioplasty
  Interventions: Procedure: Trans-inguinal Pre-peritoneal Hernioplasty
- group B (Experimental): Patients undergoing lichtnestein's hernioplasty
  Interventions: Procedure: Lichtnestein's hernioplasty

INTERVENTIONS:
Procedure: Trans-inguinal Pre-peritoneal Hernioplasty — patients were catheterised pre-operatively, to prevent any injury to the bladder and aid in preperitoneal dissection. The catheter was removed after 48 hours post-operatively.
  Incision of TIPP is same as that of Lichtenstein technique . After dissection of the sac, the transversalis is fascia is incised to enter the preperitoneal space. The preperitoneal space is developed by dissection with index finger. The space extends from rectus muscle medially, arcuate line cranially, a little beyond the anterior superior iliac spine over the psoas muscle laterally and the lilipubic tract caudally. A 15 cm x 15 cm polypropylene mesh, cut into dimension 15 cm x 12 cm, the inferior medial angle of the mesh is trimmed in a semicircular fashion to prevent trauma to the bladder neck. The mesh is placed in the preperitoneal space and anchored to the Cooper's ligament with a single 2-0 interrupted prolene suture
  Other Names: TIPP Technique
  Arms: group A
Procedure: Lichtnestein's hernioplasty — incision 1 cm above and parallel to inguinal ligament,Opening subcutaneous fat ,Opening Scarpa fascia to external oblique aponeurosis ,visualization of external ring and lower border of the inguinal ligament,Opening deep fascia of the thigh,checking for a femoral hernia ,Division of external oblique aponeurosis from external ring laterally for 5 cm, safeguarding ilioinguinal nerve ,Mobilization of superior and inferior flaps of external oblique aponeurosis exposing underlying structures ,Mobilization of spermatic cord along with the cremaster, including (ilioinguinal ,genitofemoral) nerves, and spermatic vessels; all of these structures may be encircled in a tape ,Opening of the coverings of spermatic cord, identification and isolation of the hernia sac ,Inversion, division, resection, or ligation of the sac ,Placement and fixation of mesh to edges of the defect or weakness in the posterior wall of inguinal canal creating artificial internal ring,Closure
  Arms: group B

SUMMARY:
Mesh repair of inguinal hernia is the most common operation performed on general surgical patients. Approximately 20 million groin hernioplasties are performed each year worldwide. Countless studies have been reported in the medical literature in attempts to improve the overall outcomes following hernia operations and, due to this fact, the procedure has evolved immensely, especially over the last few decades. Recurrence of inguinal hernia was initially a significant problem. Lichtenstein repair (LR), recurrence rate has consistently been reported as low as 1-4%[2], a drop from up to 10%. But increased incidence of chronic groin pain following LR.

Transinguinal preperitoneal (TIPP) inguinal hernia repair with soft mesh has been reported as a safe anterior approach with a preperitoneal mesh position .

Theoretically, TIPP repair may be associated with lesser chronic postoperative pain than Lichtenstein's technique due to the placement of mesh in the preperitoneal space to avoid direct regional nerves dissection and their exposure to bio-reactive synthetic mesh. The placement of mesh in this plane without using any suture for fixation and lack of mesh exposure to regional nerves was assumed to result in the reduced risk of developing chronic groin pain. So aim of our study to prove less hospital stay and complication and cost effectiveness for preperitoneal meshplasty

DETAILED DESCRIPTION:
This study is a prospective randomized study including all Patients with unilateral non complicated inguinal hernia who will undergo hernioplasty in surgery department at AUH during the period from 3- 2018 to 6- 2020

Methodology:

Patients will be classified into two groups according to the surgical procedure performed as follows:

* Group A: Patients undergoing TIPP hernioplasty
* Group B: Patients undergoing lichtnestein's technique hernioplasty

Sample size:15 patients for each group.

D) Exclusion criteria:

1. Patients who were unfit for operation.
2. Patients with bilateral or recurrent inguinal hernia
3. Patients aged below 18 years,
4. Patients undergoing emergency hernia repairs

ELIGIBILITY:
Inclusion Criteria:

* . Patients with unilateral non complicated inguinal hernia who will undergo hernioplasty in surgery department at AUH

Exclusion Criteria:

1. Patients who were unfit for operation.
2. Patients with bilateral or recurrent inguinal hernia
3. Patients aged below 18 years,
4. Patients undergoing emergency hernia repairs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
comparison between the 2 techniques regarding presence and duration of post-operative chronic pain | visits will be within 6 months post operative
  post operative clinical examination for assessment of the presence and duration of chronic pain

SECONDARY OUTCOMES:
Duration of hospital stay post operative | first week post operative
  comparison between the two techniques concerning Duration of hospital stay post operation after each procedure
presence of any wound complication by examining the wound | first 2 weeks post operative
  comparison between the two techniques concerning presence of any wound complications by wound examination
recurrence rate | 6 to 12 month post operative
  comparison between the two techniques concerning recurrence rate of inguinal hernia
operation time | intra-operative
  comparison between the two techniques regarding operative time
time needed for the patient to return to work | 1 month post operative
  comparison between the two techniques regarding needed time to return to work

IPD SHARING:
Plan to Share IPD: Undecided
Clinical examination will be undertaken immediately post-operative looking for any wound complication or scrotal collection .
  Clinical examination will be undertaken at 1 , 3 ,6 months post-operative looking for :-
  * Wound complication
  * Scrotal collection
  * Chronic Pain
  * Recurrence

REFERENCES:
- [Background] Cheek CM, Black NA, Devlin HB, Kingsnorth AN, Taylor RS, Watkin DF. Groin hernia surgery: a systematic review. Ann R Coll Surg Engl. 1998;80 Suppl 1:S1-80. PMID 11432408
- [Background] Heikkinen T, Bringman S, Ohtonen P, Kunelius P, Haukipuro K, Hulkko A. Five-year outcome of laparoscopic and Lichtenstein hernioplasties. Surg Endosc. 2004 Mar;18(3):518-22. doi: 10.1007/s00464-003-9119-4. Epub 2004 Jan 23. PMID 14735339
- [Background] Vironen J, Nieminen J, Eklund A, Paavolainen P. Randomized clinical trial of Lichtenstein patch or Prolene Hernia System for inguinal hernia repair. Br J Surg. 2006 Jan;93(1):33-9. doi: 10.1002/bjs.5235. PMID 16329082
- [Background] Gilbert AI, Felton LL. Infection in inguinal hernia repair considering biomaterials and antibiotics. Surg Gynecol Obstet. 1993 Aug;177(2):126-30. PMID 8251018
- [Background] Awad SS, Fagan SP. Current approaches to inguinal hernia repair. Am J Surg. 2004 Dec;188(6A Suppl):9S-16S. doi: 10.1016/j.amjsurg.2004.09.007. PMID 15610887
- [Background] Chung L, Norrie J, O'Dwyer PJ. Long-term follow-up of patients with a painless inguinal hernia from a randomized clinical trial. Br J Surg. 2011 Apr;98(4):596-9. doi: 10.1002/bjs.7355. Epub 2010 Nov 30. PMID 21656724
- [Background] Simons MP, Aufenacker T, Bay-Nielsen M, Bouillot JL, Campanelli G, Conze J, de Lange D, Fortelny R, Heikkinen T, Kingsnorth A, Kukleta J, Morales-Conde S, Nordin P, Schumpelick V, Smedberg S, Smietanski M, Weber G, Miserez M. European Hernia Society guidelines on the treatment of inguinal hernia in adult patients. Hernia. 2009 Aug;13(4):343-403. doi: 10.1007/s10029-009-0529-7. Epub 2009 Jul 28. PMID 19636493
- See also: Related Info — https://emedicine.medscape.com/article/1534281-overview
- See also: Related Info — https://emedicine.medscape.com/article/1534281-technique#c2